CLINICAL TRIAL: NCT07226349
Title: A Phase 1a/1b, Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BG-75098 Alone and in Combination With Other Agents in Patients With Advanced Solid Tumors
Brief Title: A Study of BG-75098 Alone and in Combination With Other Agents in Adults With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-75098-101; 2025-523165-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
Keywords: Cyclin-Dependent Kinase 2- Targeted Protein Degrader; CDK2; CDK4; CDK4 inhibitor
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a, Part A: Dose Escalation, BG-75098 Monotherapy (Experimental): Sequential cohorts of increasing dose levels of BG-75098 will be evaluated as monotherapy.
  Interventions: Drug: BG-75098
- Phase 1a, Part B: Dose Escalation, BG-75098 Combination (Experimental): Sequential cohorts of increasing dose levels of BG-75098 will be evaluated in combination with BGB-43395 and fulvestrant.
  Interventions: Drug: BG-75098; Drug: BGB-43395; Drug: Fulvestrant
- Phase 1b, Cohort 1: Dose Expansion, BG-75098 Combination (Experimental): Participants will receive BG-75098 at the recommended dose level from Phase 1a in combination with BGB-43395 and fulvestrant.
  Interventions: Drug: BG-75098; Drug: BGB-43395; Drug: Fulvestrant
- Phase 1b, Cohort 2: Dose Expansion, BG-75098 Monotherapy (Experimental): Participants will receive BG-75098 as monotherapy at the recommended dose level from Phase 1a.
  Interventions: Drug: BG-75098

INTERVENTIONS:
Drug: BG-75098 — Administered orally.
Drug: BGB-43395 — Administered orally.
  Arms: Phase 1a, Part B: Dose Escalation, BG-75098 Combination; Phase 1b, Cohort 1: Dose Expansion, BG-75098 Combination
Drug: Fulvestrant — Administered by intramuscular injection.
  Arms: Phase 1a, Part B: Dose Escalation, BG-75098 Combination; Phase 1b, Cohort 1: Dose Expansion, BG-75098 Combination

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BG-75098 alone and in combination with BGB-43395 and fulvestrant in participants with advanced solid tumors.

DETAILED DESCRIPTION:
This study will be conducted in 2 phases: Phase 1a Dose Escalation and Phase 1b Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have measurable disease as assessed by RECIST v1.1.
* Participants must have a stable Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Participants must have adequate organ function.
* Dose Escalation Part A: Participants with histologically or cytologically confirmed advanced, metastatic, or unresectable solid tumors potentially associated with cyclin-dependent kinase 2 (CDK2) dependency. Participants should have received prior treatment with available standard-of-care (SOC) systemic therapies for advanced/metastatic disease, or for whom standard therapy is not available or not tolerated.
* Dose Escalation Part B: Patients with histologically or cytologically confirmed advanced, metastatic, or unresectable solid tumors who have received ≥ 1 prior line of systemic therapy in the metastatic setting.
* Dose Expansion Cohort 1: Participants with histologically or cytologically confirmed advanced, metastatic, or unresectable CDK4/6 inhibitor-progressed solid tumors.
* Dose Expansion Cohort 2: Participants with advanced solid tumors. Participants with primary platinum refractory disease are not eligible. Participants should have received ≥ 1 line of platinum-containing chemotherapy and ≤ 4 prior therapeutic regimens in the advanced/metastatic setting.

Exclusion Criteria:

* For all cohorts: Prior therapy selectively targeting CDK2 inhibition or degradation.
* For combination cohorts: Prior therapy selectively targeting CDK4. Prior CDK4/6 inhibitor standard of care therapy is permitted and required in local regions where it is approved and available.
* Participants with active leptomeningeal disease or uncontrolled, untreated brain metastasis.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) | From first dose to 30 days after last dose, up to approximately 12 months
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including physical examination findings, electrocardiogram results, laboratory values, and AEs meeting protocol-defined dose-limiting toxicity (DLT) criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BG-75098 | Up to approximately 2 years
  MTD is determined based on a target for dose-limiting toxicities. MAD is defined as the maximum administered dose, and it is used when MTD is not reached.
Phase 1a: Recommended Dose(s) for Expansion (RDFE[s]) of BG-75098 as Monotherapy and in Combination with BGB-43395 and Fulvestrant | Up to approximately 2 years
  The RDFE(s) will be determined from safety, tolerability, pharmacokinetic, pharmacodynamic biomarker(s), preliminary antitumor activity, and any other relevant data that are obtained from the dose escalation phase.
Phase 1b: Objective Response Rate (ORR) as Assessed by the Investigator | Up to approximately 2 years
  ORR is defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR), as assessed by the investigator using RECIST v1.1.

SECONDARY OUTCOMES:
Phase 1a: ORR as Assessed by the Investigator | Up to approximately 2 years
  ORR is defined as the percentage of participants with best overall response of CR or PR, as assessed by the investigator using RECIST v1.1.
Phase 1a: Duration of Response (DOR) as Assessed by the Investigator | Up to approximately 2 years
  DOR is defined as the time from the first confirmed objective response assessed by the investigator using RECIST v1.1 until the first documentation of disease progression after treatment initiation or death, whichever comes first.
Phase 1a: Time to Response (TTR) as Assessed by the Investigator | Up to approximately 2 years
  TTR is defined as the time from treatment initiation to the first determination of overall response assessed by the investigator using RECIST v1.1.
Phase 1a: Progression-Free Survival (PFS) as Assessed by the Investigator | Up to approximately 2 years
  PFS is defined as the time from the date of the first dose of study treatment to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: DOR as Assessed by the Investigator | Up to approximately 2 years
  DOR is defined as the time from the first confirmed objective response assessed by the investigator using RECIST v1.1 until the first documentation of disease progression after treatment initiation or death, whichever comes first.
Phase 1b: TTR as Assessed by the Investigator | Up to approximately 2 years
  TTR is defined as the time from treatment initiation to the first determination of overall response assessed by the investigator using RECIST v1.1.
Phase 1b: Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of participants with a best overall response, of CR, PR, or stable disease assessed by the investigator using RECIST v1.1.
Phase 1b: Clinical Benefit Rate (CBR) | Up to approximately 2 years
  CBR is defined as the percentage of participants with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks.
Phase 1b: PFS | Up to approximately 2 years
  PFS is defined as the time from the date of the first dose of study treatment to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: Number of Participants with AEs | Up to approximately 2 years
  Number of participants with TEAEs and SAEs, including physical examination findings, electrocardiogram results, and laboratory values.
Observed Plasma Maximum Concentration (Cmax) of BG-75098 | Assessed at select time points between Cycle 1 and Cycle 2 (each Cycle is 28 days)
Observed Plasma Trough Concentration (Ctrough) of BG-75098 | Assessed at select time points between Cycle 1 and Cycle 2 (each Cycle is 28 days)
Area Under the Concentration-Time Curve (AUC) of BG-75098 | Assessed at select time points between Cycle 1 and Cycle 2 (each Cycle is 28 days)
Terminal Half-Life (t1/2) of BG-75098 | Assessed at select time points between Cycle 1 and Cycle 2 (each Cycle is 28 days)
Phase 1b: Plasma Concentrations of BG-75098 | Assessed at select time points between Cycle 1 and Cycle 7 (each Cycle is 28 days)
Phase 1a: Observed Plasma Maximum Concentration (Cmax) of BGB-43395 | Assessed at select time points between Cycle 1 and Cycle 2 (each Cycle is 28 days)
Phase 1a: Observed Plasma Trough Concentration (Ctrough) of BGB-43395 | Assessed at select time points between Cycle 1 and Cycle 2 (each Cycle is 28 days)
Phase 1a: Area Under the Concentration-Time Curve (AUC) of BGB-43395 | Assessed at select time points between Cycle 1 and Cycle 2 (each Cycle is 28 days)
Phase 1a: Terminal Half-Life (t1/2) of BGB-43395 | Assessed at select time points between Cycle 1 and Cycle 2 (each Cycle is 28 days)
Plasma Concentrations of BGB-43395 | Assessed at select time points between Cycle 1 and Cycle 7 (each Cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (5):
- Australia (3):
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Cabrini Hospital Malvern, Malvern East, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- Sun Yat Sen Memorial Hospital, Sun Yat Sen University (South), Guangzhou, Guangdong, China
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/